CLINICAL TRIAL: NCT01306175
Title: Relative Bioavailability of a Single Oral Dose of Digoxin (0.5 mg) When Administered Alone or in Combination With Multiple Oral Doses of BI 10773 (25 mg qd) in Healthy Male and Female Volunteers (an Open-label, Randomised, Two-way Crossover Study)
Brief Title: Drug Interaction Study of Digoxin and BI 10773
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.40; 2010-023170-40 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — Digoxin; empagliflozin

ARMS (2):
- Digoxin alone (Reference) (Experimental): Tablet, oral administration with 240 mL water
  Interventions: Drug: Digoxin
- Digoxin plus BI 10773 (Test) (Experimental): Tablets, oral administration with 240 mL water
  Interventions: Drug: Digoxin plus BI 10773

INTERVENTIONS:
Drug: Digoxin plus BI 10773 — Digoxin 0.5 mg as single dose, BI 10773 medium dose once daily
  Arms: Digoxin plus BI 10773 (Test)
Drug: Digoxin — Digoxin 0.5 mg as single dose
  Arms: Digoxin alone (Reference)

SUMMARY:
The objective of the study is to investigate the relative bioavailability of digoxin after concomitant multiple oral administration of BI 10773 and a single dose of digoxin in comparison to digoxin given alone to healthy male and female subjects.

ELIGIBILITY:
Inclusion criteria:

-Healthy male and female subjects

Exclusion criteria:

-Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.40.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Macha S, Sennewald R, Rose P, Schoene K, Pinnetti S, Woerle HJ, Broedl UC. Lack of clinically relevant drug-drug interaction between empagliflozin, a sodium glucose cotransporter 2 inhibitor, and verapamil, ramipril, or digoxin in healthy volunteers. Clin Ther. 2013 Mar;35(3):226-35. doi: 10.1016/j.clinthera.2013.02.015. PMID 23497760

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Total: This was a randomised, two-period cross-over trial, the two treatments administered were
  * A single dose of 0.5mg digoxin on day 1
  * empagliflozin (Empa) 25 mg once daily on days 1 to 8 combined with a single dose of 0.5 mg digoxin on day 5
  Between treatment periods there was a washout period of at least 14 days.
Period: First Intervention
Arm/Group | Study Total
Started | 20
Completed | 20
Not Completed | 0
Period: Washout Period of at Least 14 Days
Arm/Group | Study Total
Started | 20
Completed | 20
Not Completed | 0
Period: Second Intervention
Arm/Group | Study Total
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Total: This was a randomised, two-period, cross-over trial, the two treatments administered were
  * A single dose of digoxin 0.5 mg on day 1
  * Empagliflozin (Empa) 25 mg once daily on days 1 to 8 combined with a single dose of 0.5 mg digoxin on day 5
  Between treatment periods there was a washout period of at least 14 days.
Arm/Group | Study Total
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Digoxin: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of digoxin in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: 1.5 hours (h) prior to the first dose and 20 minutes (min), 40 min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 48h, 72h, 96h after the first dose
Population: Pharmacokinetic (PK) set comprised all evaluable subjects who took at least 1 dose of study medication with at least 1 observation for at least 1 primary PK endpoint without any important protocol violations relevant to the PK evaluation. One subject was excluded from the PK set because the pre-dose plasma concentration of digoxin was >5% of Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng-h/mL
Groups:
- Digoxin Alone: A single dose of digoxin 0.5 mg on day 1.
- Digoxin and Empa: Empagliflozin (Empa) 25 mg once daily on days 1 to 8 combined with a single dose of 0.5 mg digoxin on day 5.
Arm/Group | Digoxin Alone | Digoxin and Empa
Number analyzed (Participants) | 20 | 19
ng-h/mL | 37.8 (23.2) | 39.9 (26.0)

2. Primary Outcome: Digoxin: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of digoxin, per period.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Digoxin Alone | Digoxin and Empa
Number analyzed (Participants) | 20 | 19
ng/mL | 1.97 (43.3) | 2.25 (33.8)

3. Secondary Outcome: Digoxin: Area Under the Curve 0 to Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of digoxin in plasma over the time interval from 0 extrapolated to the time of the last quantifiable data point.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Digoxin Alone | Digoxin and Empa
Number analyzed (Participants) | 20 | 19
ng*h/mL | 24.8 (24.8) | 28.4 (24.3)

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 7 days after last administration of trial medication for Digoxin and BI 10773 + Digoxin, 30 days
Arm/Group | Digoxin Alone | Digoxin and Empa
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Digoxin Alone (N=20) | Digoxin and Empa (N=20)
Fatigue (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes